CLINICAL TRIAL: NCT03869736
Title: Evaluation of the Antidepressant Effects of Nitrous Oxide in People With Major Depressive Disorder
Brief Title: Nitrous Oxide for the Treatment of Major Depressive Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayside Health (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 438/19
Record Dates: First submitted 2018-12-16; First posted 2019-03-11 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Depression; Major Depressive Disorder
Keywords: Depression; Depressive Disorder, Major; Mood Disorders; Mental Disorders; Nitrous Oxide; Anesthetics, Inhalational; Anesthetics; Anesthetics, General; Physiologic Effects of Drugs; Analgesics, Non-Narcotic; Analgesics
MeSH Terms: conditions — Depression; Depressive Disorder, Major; Mood Disorders; Mental Disorders | interventions — Nitrous Oxide

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Nitrous Oxide 50% or 25% (Experimental): Nitrous oxide at an inhaled concentration of 50% or 25%
  Interventions: Drug: Nitrous Oxide
- Placebo (Sham Comparator): Oxygen-air mixture
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Nitrous Oxide — 1-hour sessions of inhaled nitrous oxide at concentrations of 25% or 50% (randomly assigned) to be administered weekly for 4 weeks.
  Arms: Nitrous Oxide 50% or 25%
Drug: Placebo — 1-hour sessions of inhaled oxygen-air mixture (inspired oxygen concentration ~23-30%) to be administered weekly for 4 weeks.
  Arms: Placebo

SUMMARY:
The investigators are conducting a randomized controlled trial to evaluate the antidepressant effects of nitrous oxide in people with Major Depressive Disorder (MDD). MDD is a global medical condition that causes significant health and economic burden. Recent studies have shown that a single dose of ketamine, an NMDA-antagonist, has fast and long lasting anti-depressant effect. Nitrous oxide, another NMDA-antagonist, is widely used for anesthesia and analgesia, safer to administer and has fewer side effects than ketamine.

A randomized controlled crossover feasibility study showed significant reduction in depressive symptoms at 2 and 24 hours after a single 1-hour treatment session of inhaled nitrous oxide compared with placebo. Nitrous oxide is inexpensive and can be safely administered by any trained clinician. If found to be efficacious, it could be used to provide rapid anti-depressant effect whilst the benefit of traditional anti-depressants has its delayed effect. Another potential application could be in acutely suicidal patients.

This investigated-initiated phase 2b trial will enable confirmation and extension of the findings from the feasibility study, and identify the optimal dose and regimen in a broader population of those with MDD. Participants will be randomized to receive a weekly 1-hour inhalational sessions of either nitrous oxide or placebo (oxygen-air mixture) for 4 weeks, and the nitrous group will be further randomly assigned to a dose of 50% nitrous oxide or 25% nitrous oxide. Depression severity will be assessed by a blinded observer pre-treatment and at weekly intervals during and for 4 weeks after treatment using the Hamilton Depression Rating Scale.

ELIGIBILITY:
Inclusion Criteria:

1. Adult (≥18 years, both sexes), with DSM-IV-TR criteria for MDD without psychosis, as determined using a structured clinical interview [Mini International Neuropsychiatric Interview]
2. MDD, as defined by a pretreatment score >18 on the HDRS-21 scale

Exclusion Criteria:

1. A history of bipolar disorder, schizophrenia, schizoaffective disorder, obsessive-compulsive disorder, panic disorder, or documented Axis II diagnoses; active suicidal intention, as determined by clinical interview
2. Active or recent (<12 months) substance abuse or dependence; excluding nicotine
3. Administration of NMDA-antagonists (e.g., ketamine) in previous 3 months
4. Ongoing treatment with ECT
5. Presence of acute medical illness that could interfere with study participation, including significant pulmonary disease
6. Pregnancy or breastfeeding
7. Any contraindications to the use of nitrous oxide (e.g., pneumothorax, middle ear occlusion, elevated intracranial pressure, chronic cobalamin or folate deficiency unless treated with folic acid or vitamin B12).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2019-01-22 (Actual); Primary Completion 2023-06-10 (Actual); Study Completion 2023-12-10 (Actual)

PRIMARY OUTCOMES:
Change in HDRS-21 score | over 4 weeks from baseline
  21-point Hamilton Depression Rating Scale
  Interview-based questionnaire used to measure the severity of depression. Consists of 21 items with a score calculated from the first 17 answers. Higher scores are associated with more severe depression:
  0 - 7 = Normal 8 - 13 = Mild Depression 14-18 = Moderate Depression 19 - 22 = Severe Depression > 23 = Very Severe Depression Max score = 52

SECONDARY OUTCOMES:
Treatment response and remission | at 24 hours
  Treatment response (≥50% reduction on HDRS-21) and remission (HDRS-21 ≤7 points), nitrous oxide vs. placebo
Pattern of treatment response | Up to 1 week after treatment
  Assessed using daily Profile of Mood States scale. The POMS measures six different dimensions of mood swings over a period of time. score range with lower scores indicative of people with more stable mood profiles The Profile of Mood States (POMS) questionnaire is a validated psychological test containing 65 emotions/ mood states. Participants are asked to rank their current mood states using the scale 'not at all', 'a little', 'moderately', 'quite a lot' or 'extremely'. Total Mood Disturbance (TMD) score and an analysis of tension, depression, anger, vigour, fatigue and confusion is performed based on the participants mood states. Total Mood Disturbance (TMD) can be calculated by adding the scores for Tension, Depression, Anger, Fatigue and Confusion and then subtracting the score for Vigour.
  • TMD = (Tension + Depression + Anger + Fatigue + Confusion) - Vigour
Sustainability of treatment response - change in HDRS-21 scores | over 7 weeks
  Change in the HDRS-21 score, nitrous oxide vs placebo
  HDRS-21 is an interview-based questionnaire used to measure the severity of depression. Consists of 21 items with a score calculated from the first 17 answers. Higher scores are associated with more severe depression:
  0 - 7 = Normal 8 - 13 = Mild Depression 14-18 = Moderate Depression 19 - 22 = Severe Depression > 23 = Very Severe Depression Max score = 52
Sustainability of treatment response - response and remission rates | over 7 weeks
  Response and remission rates (%), nitrous oxide vs placebo
Treatment compliance rate | over 4 weeks
  Refusal or inability to attend further treatments, nitrous oxide vs placebo
Dose effect of nitrous oxide using treatment-by-dose interaction term in a logistic regression model | over 7 weeks
  Dose effect of nitrous oxide at 25% and 50% using a treatment-by-dose (group) interaction term in a logistic regression model to assess for statistical significance.
Computerized Adaptive Test-Depression Inventory (CAT-DI) | over 7 weeks
  Adaptive testing questionnaire that assesses severity, likelihood and percentile of depression based on an average of 12 items administered from a question bank of 400 items. Questions are adapted to the participants answers and targeted to their level of impairment. Results generate include: severity of depression (normal, mild, moderate, severe), likelihood of depression (out of probability of 1), percentile of severity.
Computerized Adaptive Test-Suicide Scale (CAT-SS) | over 7 weeks
  Adaptive testing questionnaire that assesses risk and severity of suicide based on items administered from a question bank. Questions are adapted to the participants answers and targeted to their level of impairment. Results generate include: risk of suicide (low, intermediate, high) and a percentile of risk.

OTHER OUTCOMES:
Adverse events | over 7 weeks
  Psychiatric AEs, such as new suicidal ideation and psychotic symptoms Other AEs, such as cardiorespiratory AEs or nausea and vomiting

CONTACTS AND LOCATIONS:
Overall Officials: Paul Myles, MD, Principal Investigator — The Alfred
Locations (2):
- University of Chicago Medicine, Chicago, Illinois, United States
- Alfred Hospital, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No